CLINICAL TRIAL: NCT04502069
Title: Treatment of COVID-19 With Opaganib in Patients With Pneumonia Requiring Oxygen But Not Mechanical Ventilation
Brief Title: Treatment of COVID-19 With Opaganib in Patients With Pneumonia Requiring Oxygen
Acronym: Opaganib-RHB
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: To be replaced with a randomized placebo-controlled study.
Sponsor: RedHill Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABC-112
Record Dates: First submitted 2020-07-10; First posted 2020-08-06 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: COVID-19; Lung Infection
Keywords: Therapeutic Use
MeSH Terms: conditions — COVID-19 | interventions — 3-(4-chlorophenyl)-adamantane-1-carboxylic acid (pyridin-4-ylmethyl)amide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label opaganib (Experimental): opaganib dosed at 500 mg Q12 hours
  Interventions: Drug: Opaganib

INTERVENTIONS:
Drug: Opaganib — 500 mg Q12 hours orally

SUMMARY:
Patients diagnosed with COVID-19 infection will be offered treatment with Opaganib, 500 mg Q12 hours. Opaganib will be continuously administered for up to 2 weeks, until discharged on room air (if earlier than 2 weeks).

DETAILED DESCRIPTION:
Patients diagnosed with COVID-19 infection by nasopharyngeal viral swab, classified as severe disease, category 5, by the WHO Ordinal Scale For Clinical Improvement (who require oxygen support by high flow nasal cannula but do not require mechanical ventilation) at the time of initiation of therapy will be offered treatment with Opaganib, 500 mg Q12 hours.

Opaganib will be continuously administered for up to 2 weeks, until discharged on room air (if earlier than 2 weeks), upon voluntary withdrawal is initiated by the patient or when the physician decides that it is not in the patient's best interest to continue.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with proven COVID-19 infection diagnosed by nasopharyngeal viral swab who require external oxygen support by high flow nasal cannulas (HFNC) but not mechanical ventilation.
2. Pneumonia documented by chest x-ray (CXR)
3. The patient or guardian must have signed a written IRB-approved informed consent.
4. A negative pregnancy test (if woman of childbearing potential).
5. Acceptable liver and renal function:

   1. Bilirubin ≤ 1.5 times upper limit of normal (CTCAE Grade 2 baseline)
   2. AST (SGOT), ALT (SGPT) ≤ 3.0 x upper limit of normal (ULN),
   3. Serum creatinine ≤ 1.5 X ULN (CTCAE Grade 1 baseline)
6. Acceptable hematologic status:

   1. Absolute neutrophil count ≥1000 cells/mm3
   2. Platelet count ≥75,000 (plt/mm3) (CTCAE Grade 1 baseline)
   3. Hemoglobin ≥ 9 g/dL
7. Clinically acceptable blood sugar control if diabetic
8. EKG showing no QTc prolongation

Exclusion Criteria:

1. Any co-morbidity that that is considered by the treating investigator as an unacceptable risk
2. Pregnant or nursing women
3. Unwillingness or inability to comply with procedures required in this protocol.
4. Caution must be exercised in patients who are receiving drugs that were sensitive substrates of CYP450 1A2, 3A4, 2C9, 2C19 or 2D6, or strong inhibitors or inducers of all major CYP450 isozymes that cannot be stopped or replaced with another appropriate medication or not given for the duration of the clinical study. These patients must be discussed with the sponsor in order to determine appropriateness for opaganib therapy.
5. Patients who are taking warfarin, apixaban, argatroban or rivaroxaban
6. Patients with QTc prolongation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Time to breathing room air | Up to 2 weeks
  To determine the time to breathing room air (off of supplemental oxygen) after the start of opaganib treatment.
Adverse Event Grading and Coding | Up to 2 weeks
  All adverse events will be graded according to the revised NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE version 5.0). If an AE is not listed in the NCI-CTCAE v.5.0, then the Investigator will use the terms: mild, moderate, severe, life-threatening, or death to describe the maximum intensity of the AE.

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Levitt, MD, Study Director — RedHill Biopharma Limited
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No